CLINICAL TRIAL: NCT02828150
Title: Integrative Parenteral Nutrition in Hospitalized, Malnourished, Hypophagic Cancer Patients With Contraindication to Enteral Nutrition
Brief Title: Integrative Parenteral Nutrition in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015013559
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neoplasms; Parenteral Nutrition
MeSH Terms: conditions — Neoplasms; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parenteral nutrition (Experimental): Patients will receive a tailored nutritional support (parenteral nutrition) to cover estimated protein-calorie requirements
  Interventions: Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Parenteral nutrition — Patients will receive a tailored nutritional support (parenteral nutrition) to cover estimated protein-calorie requirements. Energy: resting energy expenditure [Harris-Benedict] multiplied by a factor of 1.5. Protein: 1.5 g/kg/day. In obese patients (BMI >30 kg/m2) support will be calculated on ideal body weight (BMI=23 kg/m2)

SUMMARY:
Although it is demonstrated that nutritional support can improve clinical outcomes, the literature shows that approximately 50% of cancer patients are not able to meet their estimated energy requirements. Recent clinical studies suggest that a supplementary support for parenteral nutrition (PN) could significantly help to improve the nutritional status of malnourished cancer patients.

International guidelines recommend the use of PN in malnourished, hypophagic, non-surgical cancer patients if enteral nutrition is not feasible and in patients affected by severe iatrogenic gastrointestinal complications and in whom inadequate food intake is anticipated for more than 7 days. However, there are no studies on the effects of integrative PN in hospitalized, malnourished, hypophagic, non-surgical cancer patients.

Recent studies have reported on the validity of bioelectrical impedance vector analysis in monitoring the body composition of patients receiving nutritional support. Particularly, phase angle proved to be a superior prognostic marker than other nutritional screening tools.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer (head-neck, lung, gastrointestinal, pancreas, biliary tract, haematology).
* Nutritional Risk Screening 2002 score ≥3.
* Expected duration of parenteral nutrition ≥7 days
* Availability to planned measurements
* Contraindication to enteral nutrition support
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Ongoing artificial nutrition before hospitalization
* Eastern Cooperative Oncology Group performance status >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Phase angle | 7 days
  Change in phase angle (a specific body composition parameter assessed by bioelectrical impedance vector analysis) after 7 days of nutritional support

SECONDARY OUTCOMES:
body weight | 7 days
  Change in body weight after 7 days of nutritional support
body mass index | 7 days
  Change in body mass index after 7 days of nutritional support
Handgrip strength | 7 days
  Changes in muscle strength after 7 days of nutritional support
Number of participants with treatment-related adverse events as assessed by biochemistry | 7 days
  Changes in biochemistry after 7 days of nutritional support

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caccialanza R, Cereda E, Klersy C, Bonardi C, Cappello S, Quarleri L, Turri A, Montagna E, Iacona I, Valentino F, Pedrazzoli P. Phase angle and handgrip strength are sensitive early markers of energy intake in hypophagic, non-surgical patients at nutritional risk, with contraindications to enteral nutrition. Nutrients. 2015 Mar 11;7(3):1828-40. doi: 10.3390/nu7031828. PMID 25768953